CLINICAL TRIAL: NCT01844492
Title: Improving Patient and Family Centered Care in Advanced Critical Illness
Acronym: PARTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Douglas White, MD, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO13020304
Record Dates: First submitted 2013-04-19; First posted 2013-05-01 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Anxiety; Depression
Keywords: decision making for incapacitated patients; intensive care; surrogate decision making; patient centered care; Palliative Care; End of Life; Quality of Communication
MeSH Terms: conditions — Anxiety Disorders; Depression; Death

STUDY DESIGN:
Intervention Model Description: Sample size listed is for patients (n=1420), for whom 809 surrogates completed long-term follow-up
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICU Usual Care Control (Active Comparator): described below
  Interventions: Other: ICU Usual Care Control
- The PARTNER Intervention (Experimental): described below
  Interventions: Behavioral: The PARTNER Intervention

INTERVENTIONS:
Behavioral: The PARTNER Intervention — The PARTNER intervention (PAiring Re-engineered ICU Teams with Nurse-driven Emotional Support and Relationship-building) consists of: 1) institution of a clinical pathway for family support overseen by ICU staff nurses; 2) advanced communication skills training for ICU staff nurses; 3) a multifaceted strategy to support implementation of the clinical pathway for family support.
  Arms: The PARTNER Intervention
Other: ICU Usual Care Control — The control group will receive usual care, in which the frequency and content of clinician-family communication is determined by the clinical team according to their usual practice. No study ICU has a protocolized approach to family communication and instead clinicians determine the timing and frequency of communication with families. All sites have palliative care services.
  Arms: ICU Usual Care Control

SUMMARY:
One in five deaths in the U.S. occurs in or shortly after discharge from an intensive care unit (ICU), typically following decisions made by surrogate decision makers to forego life prolonging treatment. A large body of empirical research has identified deficiencies in care processes that contribute to three important problems: 1) family members often experience poor quality communication with ICU clinicians, leading to lasting psychological distress associated with the ICU experience; 2) patients near the end of life frequently receive invasive, expensive treatment that is inconsistent with their values and preferences, and 3) end-of-life care is a major contributor to health care costs.[8, 9] Although advance care planning can prevent some unwanted treatment, many patients wish for a trial of intensive treatment when the prognosis is uncertain, and therefore it seems likely that the need for interventions to improve "in-the-moment" decisions by surrogates will persist.[10, 11]

In a pilot project, the investigators developed the PARTNER intervention (PAiring Re-engineered ICU Teams with Nurse-driven Emotional Support and Relationship-building), an interdisciplinary intervention that 1) gives new responsibilities and advanced communication skills training to existing ICU staff (local nurse leaders and social work members of the ICU team); 2) changes care "defaults" to ensure frequent clinician-family meetings; and 3) adds protocolized, nurse-administered coaching and emotional support of surrogates before and during clinician-family meetings. The objective of this proposal is to conduct a stepped wedge randomized controlled trial testing the PARTNER intervention in 5 ICUs among 1000 patients with advanced critical illness and their surrogates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Surrogate decision maker for ICU patient in one of 5 UPMC ICU's

Exclusion Criteria:

* Non-English Speaking
* Surrogate's loved one is for organ transplantation
* Not physically able to participate in family meeting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1420 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-18 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | At 6 months
  Symptom burden of anxiety and depression in family members in a telephone interview 6 months after enrollment using the validated 14-item Hospital Anxiety and Depression scale (HADS).

SECONDARY OUTCOMES:
Quality of Communication (QOC) scale | At 6 months
  Quality of communication in family members in a telephone interview 6 months after enrollment using the validated19 item Quality of Communication Scale.
Patient-and Family Centeredness of Care Scale | At 6 months
  Patient and Family -Centeredness of Care, using the 12-item Patient-Perceived Patient-Centeredness of Care Scale (PPPC) adapted for use by surrogates.
Intensive Care Unit Length of Stay | Participants will be followed for duration of ICU stay, an expected average of 21 days.
  Intensive Care Unit length of stay as assessed by abstraction of this information from hospital administrative records.
Total Hospitalization costs | Duration of hospital stay, an expected average of 4 weeks
  Total hospitalization costs by aggregating each patient's total service specific costs, generated from hospital administrative records. We will stratify this analysis by the patient's vital status at hospital discharge.
Impact of Events Scale of Care Scale | At 6 months
  We will assess symptoms of post-traumatic stress in family members in a telephone interview 6 months after enrollment using the validated 22 item Impact of Events Scale.

OTHER OUTCOMES:
Mortality | At 6 months
  Hospital mortality and 6-month mortality using hospital administrative records, and the 6-month follow-up with surrogates.
Katz Activities of Daily Living Scale | At 6 months
  Functional status of the patient using the validated Katz Activities of Daily Living Scale at 6 months.
Hospital Length of Stay | Participants will be followed for duration of hosptial stay, an expected average of 4 weeks.
  We will assess hospital length of stay.
6-month health care utilization | inclusive of index hospitalization and 6 months follow up
  We will assess patient health care utilization using hospital records and through standardized interviews with surrogates at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B. White, MD,MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Centers, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Angus DC, Barnato AE, Linde-Zwirble WT, Weissfeld LA, Watson RS, Rickert T, Rubenfeld GD; Robert Wood Johnson Foundation ICU End-Of-Life Peer Group. Use of intensive care at the end of life in the United States: an epidemiologic study. Crit Care Med. 2004 Mar;32(3):638-43. doi: 10.1097/01.ccm.0000114816.62331.08. PMID 15090940
- [Background] Prendergast TJ, Claessens MT, Luce JM. A national survey of end-of-life care for critically ill patients. Am J Respir Crit Care Med. 1998 Oct;158(4):1163-7. doi: 10.1164/ajrccm.158.4.9801108. PMID 9769276
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Wendler D, Rid A. Systematic review: the effect on surrogates of making treatment decisions for others. Ann Intern Med. 2011 Mar 1;154(5):336-46. doi: 10.7326/0003-4819-154-5-201103010-00008. PMID 21357911
- [Background] Lynn J, Teno JM, Phillips RS, Wu AW, Desbiens N, Harrold J, Claessens MT, Wenger N, Kreling B, Connors AF Jr. Perceptions by family members of the dying experience of older and seriously ill patients. SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Ann Intern Med. 1997 Jan 15;126(2):97-106. doi: 10.7326/0003-4819-126-2-199701150-00001. PMID 9005760
- [Background] Murphy DJ, Burrows D, Santilli S, Kemp AW, Tenner S, Kreling B, Teno J. The influence of the probability of survival on patients' preferences regarding cardiopulmonary resuscitation. N Engl J Med. 1994 Feb 24;330(8):545-9. doi: 10.1056/NEJM199402243300807. PMID 8302322
- [Background] Weeks JC, Cook EF, O'Day SJ, Peterson LM, Wenger N, Reding D, Harrell FE, Kussin P, Dawson NV, Connors AF Jr, Lynn J, Phillips RS. Relationship between cancer patients' predictions of prognosis and their treatment preferences. JAMA. 1998 Jun 3;279(21):1709-14. doi: 10.1001/jama.279.21.1709. PMID 9624023
- [Background] Riley GF, Lubitz JD. Long-term trends in Medicare payments in the last year of life. Health Serv Res. 2010 Apr;45(2):565-76. doi: 10.1111/j.1475-6773.2010.01082.x. Epub 2010 Feb 9. PMID 20148984
- [Background] Hogan C, Lunney J, Gabel J, Lynn J. Medicare beneficiaries' costs of care in the last year of life. Health Aff (Millwood). 2001 Jul-Aug;20(4):188-95. doi: 10.1377/hlthaff.20.4.188. PMID 11463076
- [Background] Fried TR, Bradley EH, Towle VR, Allore H. Understanding the treatment preferences of seriously ill patients. N Engl J Med. 2002 Apr 4;346(14):1061-6. doi: 10.1056/NEJMsa012528. PMID 11932474
- [Background] Sudore RL, Fried TR. Redefining the "planning" in advance care planning: preparing for end-of-life decision making. Ann Intern Med. 2010 Aug 17;153(4):256-61. doi: 10.7326/0003-4819-153-4-201008170-00008. PMID 20713793
- [Background] Schneiderman LJ, Gilmer T, Teetzel HD, Dugan DO, Blustein J, Cranford R, Briggs KB, Komatsu GI, Goodman-Crews P, Cohn F, Young EW. Effect of ethics consultations on nonbeneficial life-sustaining treatments in the intensive care setting: a randomized controlled trial. JAMA. 2003 Sep 3;290(9):1166-72. doi: 10.1001/jama.290.9.1166. PMID 12952998
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Derived] Andersen SK, Chang CH, Arnold RM, Pidro C, Darby JM, Angus DC, White DB; Pairing Re-engineered Intensive Care Teams with Nurse-driven Emotional Support, Relationship building (PARTNER) Investigators. Impact of a family support intervention on hospitalization costs and hospital readmissions among ICU patients at high risk of death or severe functional impairment. Ann Intensive Care. 2024 Jul 2;14(1):103. doi: 10.1186/s13613-024-01344-9. PMID 38954149
- [Derived] White DB, Angus DC, Shields AM, Buddadhumaruk P, Pidro C, Paner C, Chaitin E, Chang CH, Pike F, Weissfeld L, Kahn JM, Darby JM, Kowinsky A, Martin S, Arnold RM; PARTNER Investigators. A Randomized Trial of a Family-Support Intervention in Intensive Care Units. N Engl J Med. 2018 Jun 21;378(25):2365-2375. doi: 10.1056/NEJMoa1802637. Epub 2018 May 23. PMID 29791247